CLINICAL TRIAL: NCT00905333
Title: Evaluation of the Pharmacokinetic Interaction Between Candesartan and Felodipine in a Combination Package Compared to the Separate Intake of the Reference Brands Atacand and Splendil After a Fasting Period.
Brief Title: Evaluation of the Pharmacokinetic Interaction Between Candesartan and Felodipine After Ingestion of a Specific Meal
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Scentryphar Clinical Research (Other); Cori Analyticals (Unknown); Clínica São Lucas, Hospital Sírio Libanês de Itatiba S/C (Unknown); LabClin Laboratório Clínico (Unknown); Laboratório de Patologia Clínica Dr. Franceschi Ltda. (Unknown); Faculty of Pharmaceutical Sciences of Ribeirão Preto - Bioequivalence Center (Other)
Responsible Party: MC MD, AstraZeneca
Model: Crossover | Masking: None
Other Study IDs: D2452L00021; IMPACT 15381
Record Dates: First submitted 2009-05-19; First posted 2009-05-20 (Estimated); Last update posted 2010-12-07 (Estimated); Status verified 2010-12

CONDITIONS: Healthy
Keywords: pharmacokinetics; candesartan; felodipine; test formulations; Atacand®; Splendil®; healthy volunteers; blood samples; after meal intake interaction; Kinetic interaction amongst test formulations of Candesartan and Felodipine and the brands Atacand® and Splendil® in healthy volunteers after a fasting period.
MeSH Terms: interventions — candesartan; Felodipine; candesartan cilexetil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single-arm (Other): 3 treatments, 6 sequences, 3 periods, cross-over, single dose arm (Willians' Plan)
  Interventions: Drug: Candesartan (test); Drug: Felodipine (test); Drug: Candesartan Cilexetil; Drug: Felodipine

INTERVENTIONS:
Drug: Candesartan (test) — 16 mg oral tablet, single dose
Drug: Felodipine (test) — 5 mg oral extended release tablet, single dose
Drug: Candesartan Cilexetil — 16 mg oral tablet, single dose
  Other Names: Atacand®
Drug: Felodipine — 5 mg oral extended release tablet, single dose
  Other Names: Splendil®

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic interaction of test formulations of candesartan and felodipine in a combination package comparing with the fasting intake of commercial formulations of both Atacand ® and Splendil®

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* BMI > or = 19 and < or = 28 (Dietary Guidelines Advisory Committee, 2005)

Exclusion Criteria:

* Not healthy
* Chronic drug intake

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2008-10; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Kinetic interaction evaluation of two test formulations of 16 mg of candesartan and 5 mg of felodipine after a fasting period and the comparison with the intake of both reference medicaments: Atacand® and Splendil®. | 76 blood samples per subject

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Abib Junior, MD, Principal Investigator — Scentryphar Clinical Research; Moises L. P Vanuncci, MD, Study Chair — Scentryphar Clinical Research
Locations (2):
- Brazil (2):
  - Research Site, Itatiba, São Paulo
  - Research Site, Americana